CLINICAL TRIAL: NCT00000641
Title: A Phase II/III Trial of Rifampin, Ciprofloxacin, Clofazimine, Ethambutol, and Amikacin in the Treatment of Disseminated Mycobacterium Avium Infection in HIV-Infected Individuals.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 135; 11110 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Mycobacterium Avium-intracellulare Infection; HIV Infections
Keywords: Rifampin; Mycobacterium avium-intracellulare Infection; Drug Evaluation; Drug Therapy, Combination; Ethambutol; Clofazimine; Acquired Immunodeficiency Syndrome; Amikacin; Azithromycin; Ciprofloxacin
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Ciprofloxacin; Ethambutol; Amikacin; Azithromycin; Rifampin; Clofazimine

INTERVENTIONS:
Drug: Ciprofloxacin hydrochloride
Drug: Ethambutol hydrochloride
Drug: Amikacin sulfate
Drug: Azithromycin
Drug: Rifampin
Drug: Clofazimine

SUMMARY:
To compare the effectiveness and toxicity of two combination drug treatment programs for the treatment of disseminated Mycobacterium avium infection in HIV seropositive patients. [Per 03/06/92 amendment: to evaluate the efficacy of azithromycin when given in conjunction with either ethambutol or clofazimine as maintenance therapy.] Disseminated M. avium infection is the most common systemic bacterial infection complicating AIDS in the United States. The prognosis of patients with disseminated M. avium is extremely poor, particularly when it follows other opportunistic infections or is associated with anemia. Test tube studies and clinical data indicate that the best treatment program may include clofazimine, ethambutol, a rifamycin derivative, and ciprofloxacin. Test tube and animal studies indicate that amikacin is a bactericidal (bacteria destroying) drug that works better when used with ciprofloxacin. Its role in treatment programs is a key issue because of toxicity and because it must be administered parenterally (by injection or intravenously).

DETAILED DESCRIPTION:
Disseminated M. avium infection is the most common systemic bacterial infection complicating AIDS in the United States. The prognosis of patients with disseminated M. avium is extremely poor, particularly when it follows other opportunistic infections or is associated with anemia. Test tube studies and clinical data indicate that the best treatment program may include clofazimine, ethambutol, a rifamycin derivative, and ciprofloxacin. Test tube and animal studies indicate that amikacin is a bactericidal (bacteria destroying) drug that works better when used with ciprofloxacin. Its role in treatment programs is a key issue because of toxicity and because it must be administered parenterally (by injection or intravenously).

Patients undergo an initial 2-week observation period (days 1 - 14) during which time baseline evaluations are performed and type and severity of symptoms are monitored. Eligible patients are randomized on day 15 to one of two treatment programs: (1) ciprofloxacin, clofazimine, ethambutol, and rifampin (all taken orally), or (2) the same four drugs plus amikacin. Only patients for whom blood cultures obtained on either day 1 or day 14/15 are positive by week 6 continue on study drugs. Patients receive combination therapy for 24 weeks. Patients may have an indwelling central venous catheter in place for long-term administration of intravenous drug. PER 03/06/92 AMENDMENT: Newly enrolled patients who demonstrate a complete or partial clinical response at the end of study week 10 (8 weeks of drug therapy) discontinue their current regimen and begin maintenance therapy with azithromycin plus either ethambutol or clofazimine for an additional 24 weeks. Patients who do not demonstrate a response at study week 10 are discontinued from all study therapy. Patients enrolled on earlier versions of the protocol who have surpassed study week 16 (14 weeks of drug therapy) continue treatment with their originally assigned regimen through study week 26; those who have not surpassed study week 16 are considered for inclusion in the maintenance phase of the study.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Zidovudine (AZT) and didanosine (ddI). Dideoxycytidine (ddC), EPO, and other experimental therapies granted Treatment IND or Expanded Access status, with the exception of rifabutin.
* Concurrent therapies (acute and maintenance) for opportunistic infections not specifically prohibited.

Concurrent Treatment:

Allowed:

* Interferon-alfa.

Patients must have the following:

* HIV infections or diagnosis of AIDS as per CDC classification.
* Mycobacterium avium isolated from blood.
* Capability of signing an informed consent, or consent of guardian if < 18 years of age.
* Ability and willingness to participate in all components of the study and receive all study therapies.

Prior Medication:

Allowed:

* Interferon-alfa.
* Single drug prophylaxis for Mycobacterium avium or M. tuberculosis within the previous 4 weeks.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

Treatment Phase:

* Known or suspected allergy to any of the study medications. Severe hearing loss.

Maintenance Phase:

* Severe hearing loss. Hypersensitivity to macrolides. Intolerance to ethambutol and clofazimine.

Concurrent Medication:

Excluded:

* Acute therapy for other opportunistic infections at time of study entry.
* Nephrotoxic agents such as amphotericin B, intravenous vancomycin, or foscarnet during the first 4 weeks of study therapy without specific exemption from one of the protocol chairs. Antacids within 2 hours of ingestion of study drugs.
* Immunomodulators (except interferon-alfa) and other antimycobacterial drugs (including quinolones and aminoglycosides).
* All experimental therapies (except ddI, ddC, and other experimental agents granted "Treatment IND" or "expanded access" status) will be prohibited (specific exemptions must be obtained from one of the protocol chairs).

Patients with the following are excluded:

* Known or suspected allergy to any of the study medications. Cannot take drugs orally.
* Severe hearing loss, at the discretion of the investigator.

Prior Medication:

Excluded:

* Antimycobacterial drugs (including azithromycin, clarithromycin, rifamycins, quinolones, and aminoglycosides) or immunomodulators (except interferon-alfa) within 4 weeks prior to entry, except single-drug prophylaxis specifically allowed.

History of unreliable drug intake.

* Inability to cooperate in the testing procedures.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Study Completion 1994-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DM Parenti, Study Chair; J Ellner, Study Chair
Locations (16):
- United States (16):
  - Harbor-UCLA Med. Ctr. CRS, Torrance, California
  - Indiana Univ. School of Medicine, Infectious Disease Research Clinic, Indianapolis, Indiana
  - St. Louis ConnectCare, Infectious Diseases Clinic, St Louis, Missouri
  - Washington U CRS, St Louis, Missouri
  - NJ Med. School CRS, Newark, New Jersey
  - NY Univ. HIV/AIDS CRS, New York, New York
  - Beth Israel Med. Ctr. (Mt. Sinai), New York, New York
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Regional Center for Infectious Disease, Wendover Medical Center CRS, Greensboro, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - Pitt CRS, Pittsburgh, Pennsylvania
  - University of Washington AIDS CRS, Seattle, Washington

REFERENCES:
- [Background] Parent D, Ellner J, Hafner R, Williams M, Jacobs P, Hojczyk P. A phase II/III trial of Rifampin (RIF) Ciprofloxach (CIPRO), Clofazimine (CLOF), Ethambutol (ETH), +/- Amikacin (AK) in the treatment (RX) of Disseminated Mycobacterium avium (MA) infection in HIV-infected individuals (PTS). Natl Conf Hum Retroviruses Relat Infect (2nd). 1995 Jan 29-Feb 2:56
- [Background] Ellner JJ, Goldberger MJ, Parenti DM. Mycobacterium avium infection and AIDS: a therapeutic dilemma in rapid evolution. J Infect Dis. 1991 Jun;163(6):1326-35. doi: 10.1093/infdis/163.6.1326. PMID 2037799
- [Background] Parenti DM, Williams PL, Hafner R, Jacobs MR, Hojczyk P, Hooton TM, Barber TW, Simpson G, van der Horst C, Currier J, Powderly WG, Limjoco M, Ellner JJ. A phase II/III trial of antimicrobial therapy with or without amikacin in the treatment of disseminated Mycobacterium avium infection in HIV-infected individuals. AIDS Clinical Trials Group Protocol 135 Study Team. AIDS. 1998 Dec 24;12(18):2439-46. doi: 10.1097/00002030-199818000-00013. PMID 9875582